CLINICAL TRIAL: NCT04862624
Title: Efficacy of the Spanish Version of the "Catalina" Intervention Media Project and Health Study
Brief Title: Media Project and Health Study - Spanish Version
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, MarySue Heilemann, PhD, RN, FAAN, Associate Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB#19-002046
Record Dates: First submitted 2021-04-23; First posted 2021-04-28 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Depression, Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Story-based media (Experimental): Participants will receive a link to our story-based media with Latina characters.
  Interventions: Behavioral: Catalina Story-Based Web-App
- Attention control media (Active Comparator): Participants will receive a link to non-story based media that is informational and does not involve story characters.
  Interventions: Behavioral: Attention Control Web-App

INTERVENTIONS:
Behavioral: Catalina Story-Based Web-App — Latinas in the experimental group will view a story-based web-app featuring a character named "Catalina" and psycho-therapeutic modules to motivate them to take action and get help for their symptoms of depression and/or anxiety.
  Arms: Story-based media
Behavioral: Attention Control Web-App — Latinas in the attention control group will view non-story based media that is informational.
  Arms: Attention control media

SUMMARY:
We seek to test the efficacy of the Spanish version of the "Catalina" web-app intervention compared to an attention control web-app in reducing symptoms of depression and/or anxiety and motivate women to take action to get help.

ELIGIBILITY:
Inclusion Criteria:

* self identifies as Latina
* scores 10 or more on Patient Health Questionnaire-8 (PHQ-8) or General Anxiety Disorder (GAD)-7
* can read, write, and speak Spanish
* has access to the internet

Exclusion Criteria:

* currently getting treatment for depression or anxiety
* suicidal ideation identified at screening

Ages: 21 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Yes, this is determined by self report.
Enrollment: 56 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2021-11-20 (Actual); Study Completion 2021-12-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in help seeking intention and action | Baseline and 6 weeks
  Change from baseline in help seeking intentions will be assessed by the number of participants who expressed interest in, expressed intentions to take action, or reported actually taking help-seeking action (used a resource, called a clinic, made an appointment with a mental health professional, signed up for a support group, or actually attended a group or 1:1 mental health session).

SECONDARY OUTCOMES:
Change attitudes towards seeking psychological services. | Baseline and 6 weeks.
  Change in individuals' attitudes with respect to seeking psychological services will be assessed with the Inventory of Attitudes toward Seeking Mental Health Services (IASMAS). It is a 24 item scale that measures psychological openness to seeking mental health services, help seeking propensity (ability and motivation to seek help), and indifference to stigma (a person's lack of concern of what others might think of their attitude toward seeking professional help). Total scores range from 0 to 96, and higher scores indicate more positive attitudes.
Change in attitudes in mental help seeking. | Baseline and 6 weeks.
  Change in attitudes about seeking help from a mental health professional will be assessed with the Mental Help Seeking Attitudes Scale (MHSAS) which is a 9-item instrument designed to measure respondents' overall evaluation (unfavorable vs. favorable) of their seeking help from a mental health professional if they found themselves to be dealing with a mental health concern. Total scale scores range from 0 to 63, and higher scores indicate more positive attitudes toward seeking help.
Change in Anxiety | Baseline and 6 weeks.
  Change in Anxiety will be assessed by the General Anxiety Disorder 7 (GAD7) which is a self-report screening and severity measure for generalized anxiety disorder. The seven items correspond to symptoms of anxiety and are summed for a range from 0-21; a score of 10-14 indicates moderate anxiety and scores at or above 15 indicate severe anxiety
Change in Depression | Baseline and 6 weeks.
  Change in Depression will be assessed by the Patient Health Questionnaire-8 (PHQ-8) which is a self-report assessment of depression. It has been established as a valid diagnostic and severity measure. The eight items correspond to symptom-based diagnostic criteria in Diagnostic and Statistical Manual (DSM)-IV and are summed for a range from 0-24; a score of 10-14 indicates moderate depression and scores at or above 15 indicate severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: MarySue V Heilemann, PhD, RN, Principal Investigator — UCLA School of Nursing
Locations (1):
- UCLA School of Nursing, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No